CLINICAL TRIAL: NCT00776438
Title: Evaluation of the Cellular, Humoral and Mucosal Immune Response in Adults and Elderly Subjects Vaccinated Either With an Inactivated Influenza Vaccine Administered Via the Intradermal Route or an Inactivated Influenza Vaccine Administered Via the Intramuscular Route
Brief Title: Study of Immune Response in Adults and Elderly Subjects Vaccinated With Inactivated Influenza Vaccines
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GID25
Record Dates: First submitted 2008-10-17; First posted 2008-10-21 (Estimated); Last update posted 2015-06-17 (Estimated); Status verified 2015-06

CONDITIONS: Influenza; Orthomyxovirus Infections; Myxovirus Infection
Keywords: Influenza; Orthomyxoviruses; Myxovirus Infection; Inactivated Split-virion influenza vaccine; Adults; Elderly
MeSH Terms: conditions — Influenza, Human; Orthomyxoviridae Infections | interventions — Influenza Vaccines; vaxigrip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Study Group 1 (Experimental): Adult, age 18 to 40 years
  Interventions: Biological: Inactivated, split-virion, influenza vaccine
- Study Group 2 (Experimental): Adult, age 18 to 40 years
  Interventions: Biological: Inactivated, split-virion, influenza vaccine
- Study Group 3 (Experimental): Elderly, age 60 to 85 years
  Interventions: Biological: Inactivated, split-virion influenza vaccine
- Study Group 4 (Experimental): Elderly, age 60 to 85 years
  Interventions: Biological: Inactivated, split-virion influenza vaccine

INTERVENTIONS:
Biological: Inactivated, split-virion, influenza vaccine — 0.1 mL, Intradermal
  Arms: Study Group 1
Biological: Inactivated, split-virion, influenza vaccine — 0.5 mL, Intramuscular
  Other Names: Vaxigrip®
  Arms: Study Group 2
Biological: Inactivated, split-virion influenza vaccine — 0.1 mL, Intradermal
  Arms: Study Group 3
Biological: Inactivated, split-virion influenza vaccine — 0.5 mL, Intramuscular
  Other Names: Vaxigrip®
  Arms: Study Group 4

SUMMARY:
To further characterize the immune responses induced after an influenza vaccination performed either via the ID or the IM routes in two clearly distinct populations.

Objectives:

* To describe the immune response per age group and vaccine group after vaccination.
* To describe the safety of the vaccines per age group and per vaccine group after vaccination.

ELIGIBILITY:
Inclusion Criteria :

* Aged 18 to 40 years (adults) or 60 to 85 years (elderly)
* Provision of a signed informed consent
* Able to attend all scheduled visits and comply with all trial procedures
* For a woman of child-bearing potential, avoid becoming pregnant (use of an effective method of contraception or abstinence) for at least 4 weeks prior to vaccination, until 4 weeks after vaccination
* Entitlement to national social security.

Exclusion Criteria :

* For a woman of child-bearing potential, known pregnancy or positive urine pregnancy test
* Breast-feeding woman
* Participation in another clinical trial investigating a vaccine, drug, medical device or a medical procedure in the 4 weeks preceding the trial vaccination
* Planned participation in another clinical trial during the present trial period
* Known or suspected congenital or acquired immunodeficiency, immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months, or long-term systemic corticosteroids therapy
* Known systemic hypersensitivity to any of the vaccine components or history of a life-threatening reaction to the trial vaccine or to a vaccine containing any of the same substances
* Chronic illness, at a stage that could interfere with trial conduct or completion, in the opinion of the Investigator
* Current alcohol abuse or drug addiction, which may interfere with the subject's ability to comply with trial procedures
* Receipt of blood or blood-derived products in the past 3 months, which might interfere with the assessment of immune response
* Receipt of any vaccine in the 4 weeks preceding the trial vaccination
* Planned receipt of any vaccine in the 4 weeks following the trial vaccination
* Known Human Immunodeficiency Virus, Hepatitis B or Hepatitis C seropositivity
* Previous vaccination against Influenza in the previous 6 months
* Thrombocytopenia, bleeding disorder or anticoagulants in the 3 weeks preceding the inclusion contraindicating IM vaccination
* Subject deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized without his/her consent
* Febrile illness (oral temperature >=37.5°C) or moderate or severe acute illness/infection on the day of vaccination, according to investigator judgment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2007-09; Primary Completion 2009-02 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
To provide information concerning immune response to an inactivated, split-virion, influenza vaccine. | 21 days post-vaccination
To provide information concerning the safety of inactivated, split-virion, influenza vaccine. | 21 days post-vaccination and entire study duration

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sanofi Pasteur Inc
Locations (1):
- Lyon Sud, France

REFERENCES:
- [Result] Nougarede N, Bisceglia H, Rozieres A, Goujon C, Boudet F, Laurent P, Vanbervliet B, Rodet K, Hennino A, Nicolas JF. Nine mug intradermal influenza vaccine and 15 mug intramuscular influenza vaccine induce similar cellular and humoral immune responses in adults. Hum Vaccin Immunother. 2014;10(9):2713-20. doi: 10.4161/hv.29695. PMID 25483667
- See also: Related Info — http://www.sanofipasteur.com